CLINICAL TRIAL: NCT01161043
Title: An Evaluation of a New Subcutaneous Glucose Sensor in Pediatric Subjects
Brief Title: New Glucose Sensor Pediatric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CEP232
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: diabetes; glucose; sensor
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sensor (Experimental): All subjects that wear sensors (all subjects)
  Interventions: Device: Sensor wear

INTERVENTIONS:
Device: Sensor wear — All subjects to wear sensors
  Other Names: Enlite Sensor

SUMMARY:
The purpose of this study is to assess performance of a new subcutaneous glucose sensor over a seven day sensor life when used with currently marketed Medtronic Diabetes devices. In addition performance of the new sensor will be calculated for use of the new sensor with proposed new devices using new calibration algorithms.

DETAILED DESCRIPTION:
The first generation Medtronic MiniMed Subcutaneous Glucose Sensor (Sof-Sensor) was originally approved by the FDA for commercialization as part of the Continuous Glucose Monitoring System (CGMS) on June 15, 1999 (PMA 980022). The Sensor is composed of a microelectrode with a thin coating of glucose oxidase beneath several layers of biocompatible membrane. This same sensor was used as part of subsequent continuous glucose monitoring (CGM) systems, such as the Guardian REAL-Time and Paradigm REAL-Time sensor augmented insulin pump. The current configuration of sensor has undergone in vitro and in vivo testing. A new second-generation glucose sensor (herein referred to as the Comfort Sensor) has been developed. The first-generation glucose sensor was approved with reported sensor accuracy (MAD) of 18%; it was labeled for maximum use duration of 72 hours, using only the abdomen as an insertion site. The new sensor is shorter and has a smaller diameter, with a smaller gauge introducer needle. The new sensor inserter is designed to be used with the new sensor. The objectives of this study are to 1) Assess performance of the Comfort Sensor when used over a period of seven days with currently available devices, and 2) Assess performance of the Comfort Sensor when used over a period of seven days using new calibration algorithms (post-processed with algorithm for future devices). Accuracy data will be calculated based on comparing calibrated glucose sensor values to glucose meter values during in-home testing. The devices that will be used for gathering sensor data during this study will be: 1) the Comfort Sensor, 2) the MiniLink (Transmitter), and 3) the Guardian REAL-Time Display Device.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 7 through 17 inclusive
2. Diagnosed with Type 1 Diabetes Mellitus
3. Willingness to perform required study and data collection procedures and to adhere to operating requirements of the Guardian REAL-TIME System
4. Willingness to perform at least 4 capillary blood glucose tests per day while wearing the Guardian REAL-TIME System
5. Subject agrees to comply with the study protocol requirements
6. Informed Consent, Assent, HIPAA Authorization, and California Experimental Subject Bill of Rights (if applicable) signed by the subject and/or parent/guardian
7. The Subject is willing to wear the Guardian REAL-Time System for 14 days (~340 hours).

Exclusion Criteria:

1. The Subject has a history of tape allergies that have not been resolved at time of enrollment
2. The Subject has any skin abnormality (e.g. psoriasis, rash, staphylococcus infection) in the area of sensor placement that have not been resolved at the time of enrollment and would inhibit them from wearing the sensors
3. Subject has a positive pregnancy test on enrollment
4. Subject is currently participating in an investigational study (drug or device)

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Sutter Institute for Medical Research, Sacramento, California
  - Endocrinology/ University of South Florida, St. Petersburg, Florida
  - University of Minnesota Amplatz Children's Hospital, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sensor
Started | 83
Completed | 80
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- Subjects Wearing Sensors: All subjects that wear sensors (all subjects)
  Sensor wear: All subjects to wear sensors
Arm/Group | Subjects Wearing Sensors
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.5 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 44
Region of Enrollment [Number; unit: participants]
  United States | 83

OUTCOME MEASURES:

1. Primary Outcome: Glucose Sensor Accuracy When Compared to SMBG: Proportion of Glucose Sensor Readings That Met Accuracy Criteria [Time Frame: Days One Through Six of Sensor Use]
Description: The primary accuracy parameter (primary effectiveness endpoint) was the comparative readings of paired sensor and SMBG glucose readings, measured on days 1 through 6. Accuracy is defined as within 20% agreement between SMBG and paired sensor (within 20 mg/dL if SMBG ≤ 80 mg/dL). Accuracy ranges from 0 - 100, with higher number suggests better accuracy.
Time Frame: Days one through six of sensor use
Population: a total of 3496 paired sensor and SMBG readings were recorded
Measure: Mean (95% Confidence Interval); unit: % of paired SMBG/Sensor glucose values
Units Other Than Participants: paired SMBG/sensor glucose values
Arm/Group | Subjects Wearing Sensors
Number analyzed (Participants) | 83
Number analyzed (paired SMBG/sensor glucose values) | 3496
% of paired SMBG/Sensor glucose values | 72.4 [70.3 to 74.5]

2. Secondary Outcome: Device Related Moderate or Device Related Severe Adverse Events
Description: Device related moderate adverse event: low level of inconvenience or concern to the subject and may interfere with daily activities but is usually improved by simple therapeutic remedy.
  Device related severe adverse event: interrupts a subject's daily activity and typically requires intervening treatment.
  Note: device related determination is made by the site that there is a reasonable possibility that the adverse event may have been caused by the device
Time Frame: days one through six of sensor wear
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Wearing Sensors
Number analyzed (Participants) | 83
Participants | 0

ADVERSE EVENTS:
Time Frame: days one through six of sensor wear
Arm/Group | Subjects Wearing Sensors
All-Cause Mortality (participants affected / at risk) | 0/83
Serious Adverse Events (participants affected / at risk) | 0/83
Other Adverse Events (participants affected / at risk) | 0/83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days